CLINICAL TRIAL: NCT01601509
Title: Randomized Placebo-controlled Cross-over Trial of the Effect of Nasal Tramazoline With Dexamethasone in Obstructive Sleep Apnoea Patients
Brief Title: Nasal Tramazoline and Dexamethazone in Obstructive Sleep Apnea (OSA) Patients Tramazoline and
Acronym: NTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ioannis Koutsourelakis, MD, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UOA-123
Record Dates: First submitted 2012-03-04; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nasal spray with tramazoline and dexamethazone (Active Comparator)
  Interventions: Drug: Nasal tramazoline with dexamethazone
- Placebo (Placebo Comparator)
  Interventions: Drug: Nasal placebo

INTERVENTIONS:
Drug: Nasal tramazoline with dexamethazone — Every patient will undergo four assessments. Every assessment will consist of an overnight polysomnography with concomitant measurement of breathing route pattern (oral, nasal, oro-nasal breathing epochs) as previously described [7], along with a nasal resistance measurement. After baseline assessment and randomization patients of the first group will undergo a one-week therapy with nasal tramazoline and dexamethazone, while the patients of the second group will undergo a one-week therapy with nasal placebo (sodium chloride, 0.9% solution). The second assessment will take place at the end of this one week regimen. A washout period of two weeks will follow. Subsequently, the third assessment will take place and next the patients of the first group will undergo a one-week therapy with nasal placebo (sodium chloride, 0.9% solution), while the patients of the second group will undergo a one-week therapy with nasal tramazoline and dexamethazone. Fourth assessment will then follow.
  Arms: nasal spray with tramazoline and dexamethazone
Drug: Nasal placebo — Every patient will undergo four assessments. Every assessment will consist of an overnight polysomnography with concomitant measurement of breathing route pattern (oral, nasal, oro-nasal breathing epochs) as previously described [7], along with a nasal resistance measurement. After baseline assessment and randomization patients of the first group will undergo a one-week therapy with nasal tramazoline and dexamethazone, while the patients of the second group will undergo a one-week therapy with nasal placebo (sodium chloride, 0.9% solution). The second assessment will take place at the end of this one week regimen. A washout period of two weeks will follow. Subsequently, the third assessment will take place and next the patients of the first group will undergo a one-week therapy with nasal placebo (sodium chloride, 0.9% solution), while the patients of the second group will undergo a one-week therapy with nasal tramazoline and dexamethazone. Fourth assessment will then follow.
  Arms: Placebo

SUMMARY:
Nasal resistance presents considerable variations during night[8]. Additionally, Oral and oro-nasal breathing epochs exhibit strong correlation with the number of apnoea/hypopnoeas [7].The hypothesis that the present study aims to test is whether the pharmacological prevention of increased nasal resistance during night could alter breathing route pattern and lead to a decrease in the number of apnoea/hypopnoeas in OSA patients with normal nasal resistance.

DETAILED DESCRIPTION:
Nasal obstruction impairs sleep quality and may predispose to snoring and obstructive sleep apnoea (OSA) [1]. Indeed, in healthy subjects, experimental nasal occlusion has been shown to elicit obstructive apnoeas [2]. Additionally, in patients with OSA nasal obstruction is considered a risk factor for the development of OSA [3].

Despite the relationship between nasal obstruction and OSA, the therapeutic effect of improving nasal airway patency on OSA severity remains a point of conjecture [4]. In fact, administration of intranasal corticosteroids has been shown to improve sleepiness and reduce the apnoea/hypopnoea index (AHI) in patients with OSA and rhinitis [5], whereas in OSA patients with nasal obstruction the use of topical decongestants, external nasal dilators and nasal surgery has provided equivocal results [6].

The present authors have demonstrated a strong correlation between apnoea-hypopnoea index and oral/oro-nasal breathing epochs in patients with OSA and normal nasal resistance [7]. Additionally, Kohler et al [8] have shown that nasal resistance may increase during sleep reflecting substantial variability. Therefore, it is plausible to hypothesize that OSA patients presenting with normal nasal resistance when they are awake may demonstrate increased nocturnal nasal resistance during sleep that may predispose to oral/oro-nasal breathing and elicit apnoea/hypopnoeas. Prevention of nocturnal nasal obstruction in such OSA patients may decrease oral/oro-nasal breathing and eventually be beneficial for OSA by decreasing apnoea/hypopnoeas. Thus, the present study aims to investigate whether the pharmacological prevention of nasal obstruction could alter breathing route pattern and lead to a decrease in the number of apnoea/hypopnoeas in OSA patients with normal nasal resistance.

The study will include two nasal treatment options. Firstly, a combination of a nasal decongestant (tramazoline) with a nasal corticosteroid (dexamethazone). Tramazoline (imidazoline derivative) is a nasal decongestant, which attains its maximal effect between 30 and 210 min after application [9], while nasal dexamethasone can attenuate nasal inflammation associated with OSA [10]. Secondly, sodium chloride (0.9% solution).

OSA patients (AHI>10 events/h) with normal nasal resistance measured in seated and supine position with active anterior and posterior rhinomanometry (<3.0 cmH20•L-1•s) will be recruited. Exclusion criteria will be considered: 1) recent surgery involving the upper airways, 2) central apnoeas more than three per hour or five percent of total apnoeas, 3) total sleep time during polysomnographies less than three hours, 4) current treatment with nasal decongestants and topical steroids, and 5) upper or lower respiratory tract disease, including a history of nasal allergy, and 6) smoking.

A randomized double-blind, placebo-controlled, cross-over design will be used (Figure 1). Every patient will undergo four assessments which will take place 24-48 hours after each treatment arm. Every assessment will consist of an overnight polysomnography with concomitant measurement of breathing route pattern (oral, nasal, oro-nasal breathing epochs) as previously described [7], along with a nasal resistance measurement. After baseline assessment and randomization patients of the first group will undergo a one-week therapy with nasal tramazoline and dexamethazone, while the patients of the second group will undergo a one-week therapy with nasal placebo (sodium chloride, 0.9% solution). The second assessment will take place at the end of this one week regimen. A washout period of two weeks will follow. Subsequently, the third assessment will take place and next the patients of the first group will undergo a one-week therapy with nasal placebo (sodium chloride, 0.9% solution), while the patients of the second group will undergo a one-week therapy with nasal tramazoline and dexamethazone. Fourth assessment will then follow.

Figure 1. Study design

First group: one First group: one week nasal week nasal placebo tramazoline with dexamethazone

2 weeks washout period

Second group: one Second group: one week nasal placebo week nasaltramazoline with dexamethazone

First Assessment Second Assessment Third Assessment Fourth Assessment

ELIGIBILITY:
Inclusion Criteria:

1. OSA patients (AHI > 10 events/h), and
2. normal nasal resistance measured in seated and supine position with active anterior and posterior rhinomanometry (< 3.0 cmH20•L-1•s).

Exclusion Criteria:

1. recent surgery involving the upper airways,
2. central apnoeas more than three per hour or five percent of total apnoeas,
3. total sleep time during polysomnographies less than three hours,
4. current treatment with nasal decongestants and topical steroids, and
5. upper or lower respiratory tract disease, including a history of nasal allergy, and
6. smoking.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Apnoea-hypopnoea index | up to 4 weeks
  After baseline assessment and randomization first group will undergo a one-week therapy with nasal tramazoline-dexamethazone, while second group will undergo a one-week therapy with nasal placebo. The second assessment will take place at the end of one week regimen. A washout period of two weeks will follow. Subsequently, the third assessment will take place and next first group will undergo a one-week therapy with nasal placebo, while second group will undergo a one-week therapy with nasal tramazoline-dexamethazone. Fourth assessment will then follow.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Koutsourelakis, MD, Principal Investigator — University of Athens
Locations (1):
- Centre of Sleep Disorders, Athens, Greece

REFERENCES:
- [Derived] Koutsourelakis I, Minaritzoglou A, Zakynthinos G, Vagiakis E, Zakynthinos S. The effect of nasal tramazoline with dexamethasone in obstructive sleep apnoea patients. Eur Respir J. 2013 Oct;42(4):1055-63. doi: 10.1183/09031936.00142312. Epub 2013 Feb 8. PMID 23397296